CLINICAL TRIAL: NCT03589586
Title: An Open-Label Trial to Assess the Clinical Effectiveness of DermACELL AWM in Subjects With Chronic Venous Leg Ulcers
Brief Title: Clinical Effectiveness of DermACELL AWM in Subjects With Chronic Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeNet Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-18-004
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, controlled, open-label trial comparing DermACELL AWM to conventional care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DermACELL AWM + Conventional Care (Experimental): DermACELL AWM, acellular dermal matrix, plus conventional wound care- DermACELL AWM will be applied at the Baseline visit. Conventional wound care will include advanced wound dressings and multilayer compression.
  Interventions: Other: DermACELL AWM
- Conventional Care (No Intervention): Conventional wound care will include advanced wound dressings and multilayer compression.

INTERVENTIONS:
Other: DermACELL AWM — DermACELL AWM is a sterile, ready to use acellular dermal matrix
  Other Names: Acellular dermal matrix
  Arms: DermACELL AWM + Conventional Care

SUMMARY:
This study is a multicenter, randomized, controlled, open-label trial designed to evaluate the safety and efficacy of DermACELL in subjects with a single target chronic venous leg ulcer (VLU).

DETAILED DESCRIPTION:
This study is a multicenter, randomized, controlled, open-label trial designed to evaluate the safety and efficacy of DermACELL in subjects with a single target chronic venous leg ulcer (VLU). After eligibility is determined at a screening visit, VLU subjects will be entered into a 2 week run-in period of conventional wound care with moist wound therapy and multilayer compression bandage.

At baseline, those continuing to meet eligibility criteria will be randomized to either DermACELL or conventional care wound management at a ratio of 1:1. The appropriate size of DermACELL will be applied to the wound of subjects in the DermACELL arm. The ADM will be attached with sutures, sterile adhesive strips, or bioadhesive, and covered with a dressing. For subjects in the conventional care wound management arm, the debrided wound will undergo a moist-wound therapy consisting of alginates, foams, or hydrogels, and will be covered with a gauze that is appropriate for the type of wound (moist or dry).

Subsequent study visits will occur every week until 100% re-epithelialization or up to 16 weeks after treatment (whichever comes first).

ELIGIBILITY:
Inclusion Criteria:

* Have been on a stable anti-diabetic treatment for at least 30 days before the baseline visit if the subject has a diagnosis of Type 1 or Type 2 diabetes as defined by the American Diabetes Association
* Have a full-thickness venous leg ulcer that does not penetrate into the muscle, tendon or bone.
* Have a single target ulcer
* Have a wound with an area greater than or equal to 1 cm2 and less than 25 cm2 and a depth less than or equal to 9 mm
* Have a venous stasis ulcer that has been present for at least 30 days.
* Have a Clinical severity, Etiology or cause, Anatomy and Pathophysiology ulcer classification (CEAP) Grade C6: an open venous ulcer
* Have an absence of infection based on Infectious Disease Society of America criteria
* Have adequate circulation to the affected lower extremity, defined as an Ankle-brachial index (ABI) greater than 0.75.
* Have the ability to comply with off-loading (if required for specific wound), compression and dressing change requirements
* Have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by an institutional review board (IRB), and agree to abide by the study restrictions and return to the site for the required assessments
* Have provided written authorization for use and disclosure of protected health information
* Have a life expectancy of greater than 6 months

Exclusion Criteria:

* Be pregnant or lactating
* Have a venous leg ulcer on the dorsum of the foot or more than 50% of the ulcer is below the malleolus
* Have circulating hemoglobin A1c exceeding 12% within 90 days of the screening visit
* Have serum creatinine concentrations of 3.0 mg/dL or greater within 30 days prior to screening
* Have a sensitivity to either of the following antibiotics: lincomycin, gentamicin, polymyxin B, or vancomycin
* Have a sensitivity to polysorbate 20, N-lauroyl sarcosinate, benzonase or glycerol
* Have the wound treated with biomedical or topical growth factors within the previous 30 days before the screening visit
* Need for any additional concomitant dressing material other than the ones approved for this study
* Have clinical signs of an infection at the study ulcer site
* Have the inability to tolerate compression bandage
* Have a known or suspected disease of the immune system
* Have an active or untreated malignancy or active, uncontrolled connective tissue disease
* Had a treatment with immunosuppressive or chemotherapeutic agents, radiotherapy or systemic corticosteroids less than 30 days before the baseline visit
* Have presence of necrosis, purulence, or sinus tracts that cannot be removed by debridement
* Has undergone a revascularization procedure aimed at increasing blood flow in the treatment target limb less than 4 weeks before the baseline visit
* Have serum aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase levels greater than three times the normal upper limit within 30 days prior to screening
* Have active Charcot disease
* Have undergone treatment with a living skin equivalent within the last 4 weeks before the screening visit
* Have ongoing evidence of peripheral vascular disease, including greater than one nonpalpable pulse on either foot
* Have the presence of any condition that in the opinion of the investigator places the subject at undue risk or potentially jeopardizes the quality of the data to be generated

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Healing Rate | 16 Weeks
  effect of DermACELL on the proportion of chronic venous leg ulcers that have achieved 100% re-epithelialization without drainage or dressing requirements

SECONDARY OUTCOMES:
Time to wound closure | 16 Weeks
  Change in wound area over time

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Arizona Regional Medical Research, Tucson, Arizona
  - Southern Arizona VA Health Care System Department of Podiatry, Tucson, Arizona
  - Limb Preservation Platform, Fresno, California
  - LA Foot and Ankle Clinic, Los Angeles, California
  - South Florida Podiatry, Deerfield Beach, Florida
  - Doctors Research Network, South Miami, Florida
  - Purvis Moyer Foot and Ankle Center, Rocky Mount, North Carolina

IPD SHARING:
Plan to Share IPD: No